CLINICAL TRIAL: NCT06124170
Title: Evaluating the Effectiveness of Continuously Improved Pain Management in Knee Osteoarthritis-related Surgeries
Brief Title: Improved Pain Management in Knee Osteoarthritis-related Surgeries
Status: Completed | Type: Observational
Sponsor: Peng Liu (Other)
Responsible Party: Sponsor-Investigator, Peng Liu, Professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: 2023-414
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Unicompartmental Knee Arthroplasty; High Tibial Osteotomy; Pain Management
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Total knee arthroplasty (TKA): Total knee arthroplasty
  Interventions: Procedure: Preoperative pain managment; Procedure: Intraoperative pain managment; Procedure: Postoperative pain managment
- Unicompartmental knee arthroplasty (UKA): Unicompartmental knee arthroplasty
  Interventions: Procedure: Preoperative pain managment; Procedure: Intraoperative pain managment; Procedure: Postoperative pain managment
- High tibial osteotomy (HTO): High tibial osteotomy
  Interventions: Procedure: Preoperative pain managment; Procedure: Intraoperative pain managment; Procedure: Postoperative pain managment

INTERVENTIONS:
Procedure: Preoperative pain managment — propaganda and education on pain; Preemptive analgesia with celecoxib (200 mg bid) 2 days before surgery
Procedure: Intraoperative pain managment — Squeeze to expel blood (tourniquet); Before skin suture, 20 mL 0.5% ropivacaine was given subcutaneously for local infiltration anesthesia;
Procedure: Postoperative pain managment — The intravenous analgesia pump was placed until 48 h after surgery;On the second day after surgery, celecoxib (200 mg bid) was administered orally, and buprenorphine transdermal patch was applied externally until hospital discharge;FNB catheter was placed under the guidance of ultrasound and connected with an analgesic pump, the anesthesia lasted until 48 h after surgery ‡

SUMMARY:
In recent years, pain management coordinated with enhanced recovery after surgery (ERAS) has been widely applied and rapidly developed in orthopedics, showing promising prospects. Since 2016, our hospital has used a series of continuously improved pain management schemes for patients with knee OA who underwent total knee arthroplasty (TKA), unicompartmental knee arthroplasty (UKA), and high tibial osteotomy (HTO). Here, we retrospectively analyze these patients' clinical data to compare the effects of different pain intervention measures during the perioperative period on postoperative pain, functional exercise, hospital stay, and prognosis of the three surgical methods in an attempt to provide a feasible solution for pain management of these patients.

DETAILED DESCRIPTION:
We retrospectively analyzed the clinical data of patients with knee osteoarthritis (OA) who received surgical treatment to provide a feasible solution for perioperative pain management of these patients. The medical records of 714 patients with knee OA who had undergone total knee arthroplasty (n=551), unicompartmental knee arthroplasty (n=92) and high tibial osteotomy (n=71) were retrospectively analyzed and the cases were divided into Groups A, B, and C, according to the continuously optimized pain management. Clinical data including anesthesia grade, surgery time, functional exercise, hospital stay, pain, emotion, complications and prognosis were compared.

ELIGIBILITY:
Inclusion Criteria:

* first knee surgery were 50-80 years old had complete clinical and follow-up data

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status grade≥4 comorbidity with three or more systemic diseases long-term anxiety and depression, contraindications of painkillers, long-term alcoholism, or taking painkillers concomitant limb pain caused by spinal degeneration

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of 714 patients (142 men, 40 women; mean age: 38.5 years; age range: 18-64 years) with moderate or severe knee OA who had undergone TKA (n=551), UKA (n=92), or HTO (n=71) in a group of joint surgery at Sichuan Provincial People's Hospital between March 2016 and February 2022 were retrospectively analyzed. Clinical data, including age, weight, height, anesthesia grade, surgery, and time, as well as continuously improved perioperative pain management measures, were recorded.
Sampling Method: Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
visual analogue score (VAS) | 24 hours after surgery
  visual analogue score (VAS)
visual analogue score (VAS) | 72 hours after surgery
  visual analogue score (VAS)

SECONDARY OUTCOMES:
Quadriceps muscle strength | 24 hours after surgery
  Quadriceps muscle strength
Quadriceps muscle strength | 72 hours after surgery
  Quadriceps muscle strength
Scope of activities to knee joint | 24 hours after surgery
  Scope of activities to knee joint
Scope of activities to knee joint | 72 hours after surgery
  Scope of activities to knee joint

OTHER OUTCOMES:
Self-Rating Anxiety Scale (SAS) | 24 hours after surgery
  Self-Rating Anxiety Scale (SAS)
Self-Rating Anxiety Scale (SAS) | 72 hours after surgery
  Self-Rating Anxiety Scale (SAS)
Self-Rating Depression Scale (SDS) | 24 hours after surgery
  Self-Rating Depression Scale (SDS)
Self-Rating Depression Scale (SDS) | 72 hours after surgery
  Self-Rating Depression Scale (SDS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China